CLINICAL TRIAL: NCT01113697
Title: Molecular Mechanisms Involved in the Early and Late Responses to Allergen Challenge, in Asthmatic and Allergic Rhinitis Cohorts
Brief Title: Genetics of the Early and Late Response to Allergen Challenge
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Allergy, Genes and Environment Network (AllerGen) (Unknown); Networks of Centres of Excellence of Canada (Other)
Responsible Party: Principal Investigator, Scott Tebbutt, Associate Professor, University of British Columbia
Other Study IDs: H09-02114
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: allergen challenge; blood draw; gene expression analysis; protein analysis; genetics
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Clinical Investigator Collaborative (CIC) Asthma study cohort: Participants will be healthy volunteer research subjects with allergic asthma who will have an allergen inhalation challenge at CIC sites across Canada.
- Western Red Cedar Asthma study cohort: Participants will be volunteer research subjects with Western Red Cedar asthma, who will have a plicatic acid inhalation challenge at The Lung Centre at Vancouver General Hospital.
- Environmental Exposure Unit (EEU), Kingston General Hospital: Subjects will be over 19 years of age so that they qualify for studies involving allergen challenge.

SUMMARY:
The investigators are investigating the early and late responses to allergen challenge. The research participants who the investigators will study (from three cohorts) will be part of independently-approved studies involving allergen challenge. Due to the uniqueness of the cohorts for novel genetic study, it is logical that the investigators should initially undertake hypothesis-generating experiments. The investigators will obtain blood samples from the participants, both pre-challenge and post-challenge. The investigators will determine gene expression and protein differences between these samples, and investigate if there are inherited genetic differences between individuals that may predict their specific responses to allergens.

DETAILED DESCRIPTION:
Asthmatic and/or allergic rhinitis ('hay fever') individuals respond differently, but reproducibly, to allergen challenge. Some individuals develop an isolated early response while others also go on to develop a late response. In asthmatic individuals, airway narrowing represents the early phase of the asthmatic response to airway challenge; early phase onset can be detected within ten minutes of allergen inhalation, reaches a maximum within thirty minutes, and typically resolves within three hours. In 50-60% of allergic asthmatic adults, the early response is followed by the late phase asthmatic response, which usually starts between three and four hours after allergen inhalation challenge, and is characterized by cellular inflammation of the airway, increased lung tissue permeability, and mucus secretion. Thus, approximately half of allergic asthmatic subjects are 'dual responders' (developing both an early- and late-phase response following allergen inhalation challenge), 30-40% of allergic asthmatic adults develop an 'isolated early response', and <10% adults show an 'isolated late response'. In any given individual, the pattern of response is generally consistent. In allergic rhinitis individuals challenged by environmental exposure to pollen, equivalent differences exist in the proportions of subjects undergoing isolated early or dual phase nasal responses, with these responses measured by clinical end-points such as common symptoms of allergic rhinitis ('hay fever').

The role that inherited genetic variation might play in these differential early and late responses has so far been unexplored. However, recent experimental data in mouse models provide strong evidence that genetics could play an important role. When a specific intracellular pathway is disrupted by specific mouse gene-knockouts, this leads to the inhibition of a late response to allergen challenge, whilst maintaining the early response. The pathway is known as the Bcl10/Malt1 pathway, and it normally responds to allergen exposure by activating the expression of genes that code for pro-inflammatory proteins. The uncoupling of the late response from the early response suggests a possibility that genetic variation in genes involved in the human Bcl10/Malt1 pathway may influence the nature of the allergic response in humans. We will investigate whether there is a genetic basis for why some individuals develop an isolated early-phase response after allergen challenge whilst other individuals develop early- and late-phase responses (dual response).

We will recruit human allergic subjects undergoing experimentally-controlled allergen challenges. The specific airway responses of these individuals will be carefully and precisely measured, and blood samples will be collected just prior to, and two hours after, the allergen challenge. Due to the uniqueness of our cohorts for novel genetic study, it is logical that we should initially undertake hypothesis-generating experiments. Such experiments will involve the determination of differential changes in genome-wide gene expression in white blood cells and changes in the protein and lipid composition of the blood plasma, post-challenge compared to pre-challenge. We will then formulate and test hypotheses based on the results from these initial studies, as well as the specific following hypothesis: inherited genetic variation within the Bcl10/Malt1 pathway influence the early- and late-phase allergic response to allergen challenge.

Despite tremendous interest, the differences between the pathways leading to the dual response and those leading to the isolated early response are not completely understood. Understanding these differences is important for evaluating allergic diseases such as asthma and allergic rhinitis. In contrast to the more transient isolated early response, development of the late response is associated with the hallmark inflammatory features of chronic allergic disease. The combined cohorts represent a unique resource for the study of a fundamental physiologic response in allergy, and will provide genetic insight into new pathways for pharmacologic targeting in the treatment of chronic asthma and allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* participants will be healthy volunteer research subjects with allergic asthma, or
* participants will be volunteer research subjects with Western Red Cedar asthma, or
* participants will be healthy volunteer research subjects with allergic rhinitis (hay fever)
* all participants will be over 19 years of age so that they qualify for studies involving allergen challenge

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asthmatic and/or allergic rhinitis ('hay fever') individuals, 19 years or older
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2009-08; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Observational trial: Early versus Dual Asthmatic Response | 8 hours post allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Scott J. Tebbutt, Ph.D, Principal Investigator — University of British Columbia; Gail M. Bauvreau, Ph.D, Study Director — McMaster University; Anne K. Ellis, MD, Study Director — Queen's University; Christopher R. Carlsten, MD, Study Director — University of British Columbia; Danuta Radzioch, Ph.D, Study Director — McGill University
Locations (5):
- Canada (5):
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan
  - Laval University, Québec

REFERENCES:
- [Result] Kam SH, Singh A, He JQ, Ruan J, Gauvreau GM, O'Byrne PM, Fitzgerald JM, Tebbutt SJ. Peripheral blood gene expression changes during allergen inhalation challenge in atopic asthmatic individuals. J Asthma. 2012 Apr;49(3):219-26. doi: 10.3109/02770903.2011.654300. Epub 2012 Feb 9. PMID 22316092
- [Result] Singh A, Yamamoto M, Kam SH, Ruan J, Gauvreau GM, O'Byrne PM, FitzGerald JM, Schellenberg R, Boulet LP, Wojewodka G, Kanagaratham C, De Sanctis JB, Radzioch D, Tebbutt SJ. Gene-metabolite expression in blood can discriminate allergen-induced isolated early from dual asthmatic responses. PLoS One. 2013 Jul 2;8(7):e67907. doi: 10.1371/journal.pone.0067907. Print 2013. PMID 23844124
- [Result] Yang CX, Singh A, Kim YW, Conway EM, Carlsten C, Tebbutt SJ. Diagnosis of Western Red Cedar Asthma Using a Blood-based Gene Expression Biomarker Panel. Am J Respir Crit Care Med. 2017 Dec 15;196(12):1615-1617. doi: 10.1164/rccm.201608-1740LE. No abstract available. PMID 28463537
- [Result] Singh A, Shannon CP, Kim YW, Yang CX, Balshaw R, Cohen Freue GV, Gauvreau GM, FitzGerald JM, Boulet LP, O'Byrne PM, Tebbutt SJ. Novel Blood-based Transcriptional Biomarker Panels Predict the Late-Phase Asthmatic Response. Am J Respir Crit Care Med. 2018 Feb 15;197(4):450-462. doi: 10.1164/rccm.201701-0110OC. PMID 29087730